CLINICAL TRIAL: NCT00819195
Title: Anti-Inflammatory Type II Monocyte Induction by Glatiramer Acetate (Copaxone) Treatment of Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Multiple Sclerosis Society (Other); Teva Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-03877
Record Dates: First submitted 2008-12-16; First posted 2009-01-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Multiple Sclerosis
Keywords: relapsing-remitting; multiple sclerosis; Copaxone; glatiramer acetate; MS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Glatiramer Acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood mononuclear cells (PBMC) Serum RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RRMS: Relapsing-remitting multiple sclerosis patients who have not yet received glatiramer acetate (Copaxone) therapy recommended as part of clinical care
  Interventions: Drug: Glatiramer acetate
- HC: Healthy control volunteers

INTERVENTIONS:
Drug: Glatiramer acetate — 20 mg daily subcutaneous injection. Six-month duration.
  Other Names: Copaxone
  Groups: RRMS

SUMMARY:
The purpose of this study is to determine whether glatiramer acetate (Copaxone) will induce anti-inflammatory type II monocyte development during treatment of MS, and if these antigen presenting cells (APC) will promote Th2 and Treg differentiation of naïve T cells.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting (RR) MS patients (McDonald criteria)
* Ages 18-55
* Males and females
* EDSS score ≤5
* No prior treatment with Copaxone
* Prior treatment with corticosteroids or interferon-beta (-1a or -1b) is acceptable, provided there is a washout period of at least one month

Exclusion Criteria:

* Treatment with Tysabri, Novantrone or cyclophosphamide
* Treatment with other immunomodulatory therapies (e.g. imuran, mycophenolate or methotrexate)
* Primary-progressive (PP) and secondary-progressive (SP) multiple sclerosis
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Relapsing-remitting multiple sclerosis patients at the UCSF Multiple Sclerosis Center.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2008-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Production of inflammatory cytokines by monocytes and naive T cells. | 0, 1, 2, 4, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott S. Zamvil, M.D. Ph.D., Principal Investigator — UCSF Department of Neurology
Locations (1):
- UCSF Multiple Sclerosis Center, San Francisco, California, United States

REFERENCES:
- [Background] Weber MS, Prod'homme T, Youssef S, Dunn SE, Rundle CD, Lee L, Patarroyo JC, Stuve O, Sobel RA, Steinman L, Zamvil SS. Type II monocytes modulate T cell-mediated central nervous system autoimmune disease. Nat Med. 2007 Aug;13(8):935-43. doi: 10.1038/nm1620. Epub 2007 Aug 5. PMID 17676050
- [Background] Neuhaus O, Farina C, Wekerle H, Hohlfeld R. Mechanisms of action of glatiramer acetate in multiple sclerosis. Neurology. 2001 Mar 27;56(6):702-8. doi: 10.1212/wnl.56.6.702. No abstract available. PMID 11288751
- [Background] Farina C, Weber MS, Meinl E, Wekerle H, Hohlfeld R. Glatiramer acetate in multiple sclerosis: update on potential mechanisms of action. Lancet Neurol. 2005 Sep;4(9):567-75. doi: 10.1016/S1474-4422(05)70167-8. PMID 16109363
- [Background] Kim HJ, Ifergan I, Antel JP, Seguin R, Duddy M, Lapierre Y, Jalili F, Bar-Or A. Type 2 monocyte and microglia differentiation mediated by glatiramer acetate therapy in patients with multiple sclerosis. J Immunol. 2004 Jun 1;172(11):7144-53. doi: 10.4049/jimmunol.172.11.7144. PMID 15153538
- [Background] Weber MS, Starck M, Wagenpfeil S, Meinl E, Hohlfeld R, Farina C. Multiple sclerosis: glatiramer acetate inhibits monocyte reactivity in vitro and in vivo. Brain. 2004 Jun;127(Pt 6):1370-8. doi: 10.1093/brain/awh163. Epub 2004 Apr 16. PMID 15090474